CLINICAL TRIAL: NCT02857075
Title: Enlargement of the SmarTTransfuser Biochip (ABO Compatibility) to the Detection of Rhesus (RH1)
Brief Title: Development a Rhesus Type Compatibility Test by Means of an Antibody Able to Recognize RH1 Antigen Grafted on a Biochip
Acronym: ABORDAGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2013/38
Record Dates: First submitted 2016-07-25; First posted 2016-08-05 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Rh Incompatibility Reaction
MeSH Terms: interventions — Blood Donation

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rhesus positive individuals: Red cell concentrates from RH1 individuals from each ABO group is used for the study. Red cell concentrates derived from blood donation.
  Interventions: Other: Blood donation
- Rhesus negative individuals: red cell concentrates from RH-1 individuals from each ABO group is used for the study. Red cell concentrates derived from blood donation.
  Interventions: Other: Blood donation

INTERVENTIONS:
Other: Blood donation — Red cell concentrates derived from healthy blood donating people. In France, all blood donation is realized by the Etablissement Français du Sang, so all the study samples are from this center.

SUMMARY:
Every year, several millions of red cell concentrates are transfused. For each of them, a pretransfusional compatibility test is performed. In France, an ABO compatibility test at the patient's bedside is performed, but rhesus compatibility is not yet checked. However, rhesus antigens are very immunogenic and could lead to Rh incompatibility or Rh disease.

The objective of ABORDAGE project is to develop another biochip that specifically captures RBCs according the presence of the RH1 antigen (also known as D antigen) at their surface.

DETAILED DESCRIPTION:
Every year, several millions of red cell concentrates are transfused. For each of them, a pretransfusional compatibility test is performed. In France, an ABO compatibility test at the patient's bedside is performed, but rhesus compatibility is not yet checked. However, rhesus antigens are very immunogenic and could lead to Rh incompatibility or Rh disease. Rh incompatibility occurs when a woman with Rh-negative blood type is exposed to Rh-positive blood cells. This exposure leads to the sensitization of the women who develop anti-Rh immunoglobulin G (IgG). This immunization is one cause of the hemolytic disease of newborns (HDN). HDN results from an incompatibility between mother's blood and fetus' blood. It happens when fetal red blood cells (RBCs) present antigens inherited from the father but missing from the mother. Consequence of this incompatibility is the fetal RBCs destruction by mother's antibodies. Antibodies could be natural, like immunoglobulin M (IgM) anti-A or anti-B from the ABO system, or from an immunization. Rh incompatibility results from 2 main mechanisms. The first one is when a pregnancy Rh-negative woman is exposed to fetal Rh-positive RBCs. Rh incompatibility leads to anemia (mild to severe) or ultimately to the in utero death. The second occurs when Rh incompatible blood is transfused. This is the subject of this communication.

The investigators previously develop biochips and optical device to realize automatic ABO compatibility test at the patient's bedside (references to the Citation field). Based on this previously project, the goal of ABORDAGE project is to develop another biochip based on selective blood capture. The ABORDAGE chip has to specifically capture RBCs according the presence of the RH1 antigen (also known as D antigen) at their surface.

ELIGIBILITY:
Inclusion Criteria:

* Donor inclusion criteria will be those of the Etablissement Français du Sang

Exclusion Criteria:

* Donor exclusion criteria will be those of the Etablissement Français du Sang

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: RH1 and RH-1 red cell concentrates, derived from blood donation, is used for this study
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Detection of presence or absence of red blood cell on biochips by measurement of optical absorption with a detection module. | between 6 and 42 days after blood donation
  Detection of red blood cell capture relies on optical absorption. Electroluminescent diodes will illuminate the surfaces of biochips and photoreceptors placed opposite will detect the amount of light which crosses the surfaces. First, a reference value is taken. Then, blood is injected on the surface and rinsed, to remove unbound ligands. If red blood cells have been trapped, light is absorbed. If not, no absorption is observe.
  Absorbance level are collected and correlation between the percentage of red cells on surfaces and absorbance are analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Wacogne, PhD, Principal Investigator — CHRU besancon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charrière, K., A. Rouleau, O. Gaiffe, J. Fertey, P. Morel, V. Bourcier, C. Pieralli, W. Boireau, L. Pazart, and B. Wacogne. 2015. "Biochip Technology Applied to an Automated ABO Compatibility Test at the Patient Bedside." Sensors and Actuators B: Chemical 208 (March): 67-74. doi:10.1016/j.snb.2014.10.123.
- [Background] Charrière, Karine, Alain Rouleau, Olivier Gaiffe, Pascal Morel, Véronique Bourcier, Christian Pieralli, Wilfrid Boireau, Lionel Pazart, and Bruno Wacogne. 2015. "An Automated Medical Device for Ultimate ABO Compatibility Test at the Patient's Bedside - Towards the Automation of Point-of-Care Transfusion Safety:" In , 58-67. Lisbon, Portugal: SCITEPRESS - Science and and Technology Publications. doi:10.5220/0005248700580067.